CLINICAL TRIAL: NCT03488979
Title: Effect of Providing Education and Patient's Inferior Vena Cava Ultrasound Images on Adherence to a Heart Failure Regimen
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00034300
Record Dates: First submitted 2018-02-16; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Heart Failure; Medication Adherence
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Educational Interventional Group: Primary outcome measure: Difference in MOSSAS-3HF score between intervention group and control group, administered 4 weeks after discharge.
  Interventions: Other: educational interventional group
- Attention Control Group: Primary outcome measure: Difference in MOSSAS-3HF score between intervention group and control group, administered 4 weeks after discharge.

INTERVENTIONS:
Other: educational interventional group — • Patient Education Tool (Appendix 3) and the patient's own IVC images will be shared with each patient in the intervention group in real time. If feasible, each intervention patient will also receive a printed copy of his or her IVC image.
  Groups: Educational Interventional Group

SUMMARY:
Heart failure is a common, costly, and disabling condition characterized by recurrent exacerbations. Episodes of acute decompensated heart failure (ADHF) account for the largest proportion of admissions and 30-day readmissions to US hospitals. Medication nonadherence and dietary/fluid nonadherence have been associated with re-admissions. Hand-carried ultrasound (HCU) devices are portable, relatively inexpensive, and can augment the physical exam in the assessment of volume status. Dilated Inferior Vena Cava (IVC) with poor collapsibility correlates with elevated central venous pressure, which may be correlated with earlier readmission for ADHF.

Study design to measure maximum IVC diameter (IVC max) in mm and the degree of IVC collapsibility with inspiration on qualitative assessment in approximately 100 patients admitted with ADHF. The co-investigator will share the IVC images and interpretation with educational intervention group patients in real time; IVC images and interpretation will not be shared with control group patients. Study team will assess whether sharing these IVC measurements correlates with greater adherence to heart failure self-management after discharge, as measured by the administration of the Medical Outcomes Study Specific Adherence Scale, modified to a 3-item version relevant for patients with heart failure (MOSSAS-3HF) at 4 weeks after discharge. Study team will also assess for any difference in 30-day readmission rates for intervention vs. control group patients.

DETAILED DESCRIPTION:
The following list indicates the sequence and timing of our study procedures:

* Inpatients will be screened for study eligibility by one of the co-investigators via review of the electronic medical record (EMR) for administration of intravenous (IV) diuretics and documentation of acute decompensated heart failure (ADHF) as the indication for diuresis.
* Eligible patients will be invited to participate by a research assistant.
* All consenting patients' demographic data will be recorded. A Study Identification Number will be assigned and personal identifiers will be logged in a "key" separate from the dataset. The number of subjects who are approached but decline enrollment will be documented.
* Baseline adherence to heart failure self-management regimen will be assessed by administration of the Medical Outcomes Study Specific Adherence Scale, a 3-item questionnaire for patients with heart failure (MOSSAS-3HF). The 3 questions in the MOSSAS-3HF ask patients to rate how often in the past 4 weeks they adhered to their medication regimen, low-salt diet, and daily weight measurement. Answer choices for each of the 3 items range from 0 (none of the time) to 5 (all of the time), so a maximum total score would be 15, for adherence "all of the time" to each of the 3 items. Baseline health beliefs regarding benefits of treatments for heart failure and self-efficacy will be assessed.
* Patients who consent will be randomized into attention control group or educational intervention group using sealed envelopes (randomization generated in sets of 6 for a total of one hundred participants by using Research Randomizer).
* All participants will undergo a limited bedside HCU examination of the inferior vena cava.
* A patient education tool and the patient's own IVC images will be shared with each patient in the intervention group in real time.
* All images will be acquired by an experienced registered board certified ultrasonographer between 36 and 60 hours after admission using an HCU device by Sonosite®.
* Each HCU examination is estimated to last 3-10 minutes. All IVC studies will be performed with the patient in the supine position using the HCU machine (Sonosite Inc., Washington). Ultrasound probe will be at subxyphoid placement. Measurements will be taken using 2-D images at approximately 2 cm from the IVC/right atrium juncture, taking care to avoid any hepatic veins emptying into the IVC at the approximation of IVC/ right atrium interface. The IVC normally collapses with inspiration and expands with expiration. For this reason, patients may be asked to "sniff" to measure IVC collapsibility with inspiration.
* For patients under isolation precautions, standard hospital disinfectant procedures as recommended by the manufacturer and as followed by echocardiography department will be followed.
* The ultrasonographer will calculate and document the patient's IVC max and qualitative Inferior Vena Cava Collapsibility Index (IVCCI).
* Two weeks after discharge, a follow up phone call will be made to the all participants. The scripted phone call for intervention patients will reinforce heart failure self-management education from the Patient Education Tool. The scripted phone call for control patients will only ask neutral questions about progress since hospital discharge and whether the patient remembers getting an ultrasound in the hospital as part of the research study.
* A phone call will be made and a letter will be mailed to the participants approximately 3 weeks after the study enrollment date to serve as a reminder for the final 30-day phone call.
* A research assistant will contact all enrolled patients by telephone 4 weeks after discharge to administer MOSSAS-3HF and to ask whether the patient required hospital admission or emergency department care since the original hospital discharge where patient was enrolled in the study.
* Review of electronic medical records will be used to determine length of stay and whether patients were readmitted to Johns Hopkins Bayview Medical Center or Johns Hopkins Hospital within 30 days; for those patients not readmitted within 30 days, an attempt will be made to determine whether the patient has been readmitted to another hospital or sought care at another Emergency Department during the follow up telephone call.
* All HCU examinations will be recorded and available for review by a board-certified cardiologist.
* If an enrolled patient requests termination of the HCU examination at any time, it will stop immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized on the general inpatient medicine service
* Receiving intravenous diuretics for treatment of acute decompensated heart failure

Exclusion Criteria:

* Pregnancy
* Inability or unwillingness to provide informed consent
* Inability to read or speak English
* Without access to a working telephone number
* Recent abdominal surgery or current symptom of severe abdominal pain that would interfere with patient tolerance of pressure from an ultrasound probe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, non-pregnant patients admitted on a general inpatient medicine service of an urban, academic medical center, receiving intravenous diuretics for the treatment of acute decompensated heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
MOSSAS-3HF score | 30 days after hospital discharge
  The MOSSAS-3HF instrument is a 3-item questionnaire that assesses patient self-reported adherence to a heart failure treatment regimen over the past 4 weeks. Minimum score is 0 (adherence none of the time) and maximum score is 15 (adherence all of the time).

SECONDARY OUTCOMES:
survival without need for acute medical care within 30 days | 30 days after discharge
  assessed by scripted post-discharge telephone call
survival without need for acute medical care within 30 days | 30 days after discharge
  as assessed by review of electronic medical records

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzgerald AA, Powers JD, Ho PM, Maddox TM, Peterson PN, Allen LA, Masoudi FA, Magid DJ, Havranek EP. Impact of medication nonadherence on hospitalizations and mortality in heart failure. J Card Fail. 2011 Aug;17(8):664-9. doi: 10.1016/j.cardfail.2011.04.011. Epub 2011 Jun 23. PMID 21807328
- [Background] Martin LD, Howell EE, Ziegelstein RC, Martire C, Whiting-O'Keefe QE, Shapiro EP, Hellmann DB. Hand-carried ultrasound performed by hospitalists: does it improve the cardiac physical examination? Am J Med. 2009 Jan;122(1):35-41. doi: 10.1016/j.amjmed.2008.07.022. PMID 19114170
- [Background] Goonewardena SN, Gemignani A, Ronan A, Vasaiwala S, Blair J, Brennan JM, Shah DP, Spencer KT. Comparison of hand-carried ultrasound assessment of the inferior vena cava and N-terminal pro-brain natriuretic peptide for predicting readmission after hospitalization for acute decompensated heart failure. JACC Cardiovasc Imaging. 2008 Sep;1(5):595-601. doi: 10.1016/j.jcmg.2008.06.005. PMID 19356487
- [Background] Parkes G, Greenhalgh T, Griffin M, Dent R. Effect on smoking quit rate of telling patients their lung age: the Step2quit randomised controlled trial. BMJ. 2008 Mar 15;336(7644):598-600. doi: 10.1136/bmj.39503.582396.25. Epub 2008 Mar 6. PMID 18326503
- [Background] Spencer KT, Anderson AS, Bhargava A, Bales AC, Sorrentino M, Furlong K, Lang RM. Physician-performed point-of-care echocardiography using a laptop platform compared with physical examination in the cardiovascular patient. J Am Coll Cardiol. 2001 Jun 15;37(8):2013-8. doi: 10.1016/s0735-1097(01)01288-8. PMID 11419879
- [Background] Decara JM, Kirkpatrick JN, Spencer KT, Ward RP, Kasza K, Furlong K, Lang RM. Use of hand-carried ultrasound devices to augment the accuracy of medical student bedside cardiac diagnoses. J Am Soc Echocardiogr. 2005 Mar;18(3):257-63. doi: 10.1016/j.echo.2004.11.015. PMID 15746716